CLINICAL TRIAL: NCT04294173
Title: Effect Of Video Based Teaching On Nursing StudentsTracheostomy Care Skills
Brief Title: The Effect Of Video Based Teaching On Tracheostomy Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Seda CEVHEROĞLU, PhD Student of Nursing / Senior Instructor Department of Nursing Faculty of Health Sciences, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DAU-NURSING
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Skill, Coping; Satisfaction; Anxiety
Keywords: tracheostomy care; video training; demonstration; nursing student
MeSH Terms: conditions — Personal Satisfaction; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video group (Experimental): Within the scope of Nursing Fundamentals course, a 4-hour theoretical training will be given to the experimental group in the classroom setting. Video presentation including powerpoint presentation and tracheostomy care skill application will be prepared in line with the Respiratory System course content. The powerpoint presentation prepared will be explained by the researchers to the video group students in the classroom by question, answer, discussion and demonstration methods. Immediately after the lecture, students will be watched by the video-assisted teaching method, and the video of tracheostomy care The videos will be sent to students via e-mail. A two-day warning message will be sent to the students from the WhatsApp group to watch the video by the researchers. A week later, students will be invited to the basic skills laboratory for tracheostomy care.
  Interventions: Behavioral: video education
- demonstration group (No Intervention): Within the scope of Nursing Fundamentals course, a 4-hour theoretical training will be given to the control group in the classroom setting. Powerpoint presentation will be prepared in line with the Respiratory System course content. The powerpoint presentation prepared will be explained to the control group students by the researchers in the classroom by question, answer, discussion and demonstration methods. Immediately after the lecture, students will be taken to the basic skills laboratory and tracheostomy care will be performed on the dummy by the researchers using the demonstration method. Then, students will be given the output of the powerpoint presentation and asked to study the lecture notes for a week. A two-day warning message will be sent by the researchers to students from the WhatsApp group to study. A week later, students will be invited to the basic skills laboratory to practice tracheostomy care.

INTERVENTIONS:
Behavioral: video education — tracheostomy care will be given to student nurses with video training
  Arms: video group

SUMMARY:
The aim of this study is to evaluate the effect of video assisted instruction on nursing students' tracheostomy care skills.

The universe of the research consists of 81 students who enrolled in the Eastern Mediterranean University Faculty of Health Sciences Nursing Undergraduate Program in the fall semester of the 2019-2020 academic year and enrolled in the nursing principles course. Students who will not participate in the sample selection, agree to participate in the study voluntarily and meet the inclusion criteria, constituted the sample of the study. The research was designed on two groups, the video-based teaching method-based education (initiative) group and the demonstration (control) group. The students were divided into two randomized groups as intervention and control groups by using random numbers table.

Personal Data Form, Tracheostomy Care Skill Assessment Form, Satisfaction from Training Methods and State-Trait Anxiety Inventory were used to collect the data.

DETAILED DESCRIPTION:
Nursing education is an education system structured in order to provide the student with a professional nursing identity and to prepare the student for professional life, where theoretical and practical education is offered as a whole. In this system, nursing students are expected to acquire cognitive, affective and psychomotor skills at a very good level. Teaching process of psychomotor skill; It enables students to practice, analyze and develop skills by analyzing the theoretical information they have learned, to establish a relationship between theory and practice, to develop critical thinking and problem solving skills, to make regular observations and to gain a sense of trust . Today, with the development of technology and changing needs, there are also changes in the methods of education and training commonly used. One of the educational methods developed with technology is the video model method. Videos are among the important technologies that add value to the learning content. The use of video helps students learn new skills and improve their learning processes in the same way they have experience during practical training . Using videos while teaching nursing skills is as effective as demonstration as it provides visuality. Using a properly formatted video to teach a particular nursing skill allows a student to learn physical action that complements the theory behind skill and action. The use of training based on the video model method is useful for applications of nursing skills based on flexibility and capacity for students to review, reflect and repeat recordings . When the studies using video method in nursing education are examined; Lee et al. (2016) first shot a urinary catheterization skill video to teach nursing second grade students about urinary catheterization skills. Later, the experimental group (n = 36) was trained by mobile-based video learning and the control group students (n = 35) by the demonstration method. All students attended a 90-minute course on urinary catheterization and all students watched the urinary catheterization skill video. Students in the control group only watched the one-time video, students in the experimental group had the opportunity to watch the video for seven days on their mobile devices. A week later, students in the experimental and control groups performed urinary catheterization skill in the skill laboratory. At the end of the application, students' learning motivation, skill performance score, application confidence and skill laboratory satisfaction were evaluated. It was found that students in the experimental group had higher motivation to learn, skill laboratory satisfaction, knowledge and skill performance score and application confidence compared to the control group . Gowri, Minolin and Thenmozhi (2013) conducted a semi-experimental study in order to teach obstetric palpation skills to nursing second year students in antenatal period.

ELIGIBILITY:
Inclusion criteria:

* Being volunteer to participate in the research
* Taking the fundamentals of nursing for the first time
* No clinical experience

Exclusion criteria:

* Being the second time of nursing basis course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Tracheostomy Care Ability | 1 month
  The literature was scanned and tracheostomy care skill assessment guide was prepared by the researchers. This guidebook is a 32-item form of the procedure for preparing the psychomotor skill levels of the students in the video and demonstration group regarding the care of the patient with tracheostomy. While evaluating the forms, the observed steps will be divided into "full" and "incorrect", 1 point will be given for the fully applied step and 0 points will be given for the wrongly applied and not observed steps. Every correct step applied by students is calculated as "1" point, and every step that is not done or wrong is calculated as "0" point. The minimum score obtained from the Tracheostomy Care Skill Evaluation Form is 32 and the maximum score is 0. The skill assessment form prepared was presented to the opinion of three faculty members who are experts in the field of nursing principles in terms of scope validity.
Continuity-Status Anxiety Level | 1 month
  The Inventory is composed of two parts: State Anxiety Inventory and Trait Anxiety Inventory. In the State Anxiety Inventory, the individual needs to be able to express how he feels under certain conditions, and in the Trait Anxiety Inventory, he usually needs to express how the individual feels. The big score from the scales expresses the high anxiety level, the small score indicates the low anxiety level. He states that 0-19 points obtained from the State-Trait Anxiety Inventory are not anxiety, 20-39 points mean mild, 40-59 points mean moderate, 60-79 points mean severe anxiety, and individuals who score 60 or more need professional help.
Level Of Satisfaction FromEducation Methods | 1 month
  The survey consists of 16 propositions. One of these propositions is the proposition "I am satisfied with this training method in general", which questions the satisfaction with education. Other propositions, on the other hand, are composed of propositions aimed at determining the opinions of the education method about the contribution of the student to learning and professional life. Each proposition is scored on the 5-point Likert scale. It is determined that as the scale score increases, the satisfaction of the students from the education method increases, and as the scale point average decreases, their satisfaction from the education method decreases. In the evaluation of the scale, a minimum of 16 and a maximum of 80 points are given to the satisfaction of the students with the education methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean Unıversıty, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee NJ, Chae SM, Kim H, Lee JH, Min HJ, Park DE. Mobile-Based Video Learning Outcomes in Clinical Nursing Skill Education: A Randomized Controlled Trial. Comput Inform Nurs. 2016 Jan;34(1):8-16. doi: 10.1097/CIN.0000000000000183. PMID 26389858
- [Result] Salina L, Ruffinengo C, Garrino L, Massariello P, Charrier L, Martin B, Favale MS, Dimonte V. Effectiveness of an educational video as an instrument to refresh and reinforce the learning of a nursing technique: a randomized controlled trial. Perspect Med Educ. 2012 May;1(2):67-75. doi: 10.1007/s40037-012-0013-4. Epub 2012 Apr 28. PMID 23316461